CLINICAL TRIAL: NCT00730821
Title: A Combination Phase I Open Label Dose Escalation Study of Concomitant Administration of BIBW 2992 With BIBF 1120 in Patients With Advanced Solid Tumors
Brief Title: Phase I of BIBW 2992/BIBF 1120 Combination Therapy in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Purpose: Treatment
Other Study IDs: 1239.1
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib; nintedanib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: BIBW 2992; Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBW 2992
Drug: BIBF 1120

SUMMARY:
The primary objective of this trial is to determine the MTD of the combination of BIBW 2992/BIBF 1120 therapy administered concomitantly in a 28-day cycle schedule.

Secondary objectives are the collection of antitumor efficacy data, the determination of pharmacokinetic parameters of BIBF 1120 and BIBW 2992, and if data allow the determination of the pharmacokinetic influence of BIBW 2992 on BIBF 1120 and vice versa.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with confirmed diagnosis of advanced, non-resectable and/or metastatic solid tumors, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment.
2. Age 18 years or older.
3. Life expectancy of at least three (3) months.
4. Written informed consent that is consistent with ICH-GCP guidelines.
5. Eastern Cooperative Oncology Group performance score 0, 1or 2.
6. Patients recovered from any therapy-related toxicities from previous chemo-,hormone-, immuno-, or radiotherapies to CTC <= Grade 1.
7. Patients must have recovered from previous surgery.

Exclusion Criteria:

1. Active infectious disease.
2. Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea.
3. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol.
4. Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least four (4) weeks, no history of cerebral edema or bleeding in the past four (4) weeks and no requirement for steroids or anti-epileptic therapy.
5. Cardiac left ventricular function with resting ejection fraction <50%.
6. Absolute neutrophil count (ANC) less than 1500/mm3.
7. Platelet count less than 100,000/mm3.
8. Bilirubin greater than 1.5 mg/dl (>26 ¿mol /L, SI unit equivalent).
9. Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than two and a half times the upper limit of normal (2.5 X ULN ).
10. Serum creatinine greater than 1.5 mg/dl (>132 ¿mol/L, SI unit equivalent).
11. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception.
12. Pregnancy or breast-feeding.
13. Treatment with other investigational drugs; chemotherapy, immunotherapy, radiotherapy or hormone therapy (including LHRH agonists, megestrol acetate, or other hormones taken for breast cancer or prostate cancer); participation in another clinical study within the past 4 weeks before start of therapy or concomitantly with this study. Treatment with bisphosphonates is allowed.
14. Treatment with an EGFR- or HER2 inhibiting drug within the past 4 weeks before start of therapy or concomitantly with this study (2 weeks for trastuzumab).
15. Patients unable to comply with the protocol.
16. Active alcohol or drug abuse.
17. Patients who require therapeutic anticoagulation or antiplatelet therapy [except treatment with Aspirin (Acetylsalicylic Acid)].
18. Patients with history of haemorrhagic or thrombotic events (including transient ischemic attacks) in the past 12 months. Known inherited predisposition to bleeding or thrombosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this trial is the safety of the combination of BIBW 2992/BIBF 1120 when administered concomitantly, and this is assessed by the dose limiting toxicity | Until undue toxicity or progressive disease.

SECONDARY OUTCOMES:
Pharmacokinetics, Objective tumor response. | Until undue toxicity or progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- United States (4):
  - 1239.1.3 Boehringer Ingelheim Investigational Site, Scottsdale, Arizona
  - 1239.1.1 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1239.1.2 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1239.1.4 Boehringer Ingelheim Investigational Site, Omaha, Nebraska